CLINICAL TRIAL: NCT06285760
Title: SANDI STUDY: Effect of Acetazolamide on Diuresis and Natriuresis in Patients With Acute Heart Failure.
Brief Title: Effect of Acetazolamide on Diuresis and Natriuresis in Patients With Acute Heart Failure (SANDI STUDY)
Acronym: SANDI
Status: Recruiting | Type: Observational
Sponsor: Puerta de Hierro University Hospital (Other)
Collaborators: Hospital Clinic of Barcelona (Other); Hospital Central de la Defensa Gómez Ulla (Other); Hospital Vall d'Hebron (Other); Hospital Universitario Ramon y Cajal (Other); University Hospital of Girona Dr. Josep Trueta (Network); Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other)
Responsible Party: Principal Investigator, Julia Gonzalez, Cardiologist, Puerta de Hierro University Hospital
Other Study IDs: 135/23
Record Dates: First submitted 2024-01-08; First posted 2024-02-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Heart Failure; Persistent Congestion
Keywords: Acetazolamide
MeSH Terms: conditions — Heart Failure | interventions — Acetazolamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Hospitalized heart failure patients: Patients hospitalized with decompensated heart failure and fluid overload who require diuretic treatment for relieve of congestion. Standarized diuretic protocol according to guidelines will be applied, including loop diuretic and sodium-glucose cotransporter-2 inhibitors (SGLT2i)
  Interventions: Drug: Acetazolamide 500mg

INTERVENTIONS:
Drug: Acetazolamide 500mg — Patients hospitalized with decompensated heart failure and fluid overload who require diuretic treatment for relieve of congestion. Standarized diuretic protocol according to guidelines will be applied. It consists of intravenous furosemide, SGLT2 inhibitors and acetazolamide if congestion persist.

SUMMARY:
The goal of this observational study is to assess the natriuretic effect of intravenous acetazolamide in patients admitted with heart failure and persistent congestion despite treatment with intravenous furosemide and sodium-glucose cotransporter type 2 (iSGLT2) inhibitors.

The main question it aims to answer is whether there is a difference in natriuresis 24 hours after acetazolamide association to medical treatment recommended by the guidelines (furosemide and ISGLT2).

DETAILED DESCRIPTION:
The SANDY study is a prospective, multicenter, observational study that will be conducted across 11 hospitals in Spain. It will enroll patients hospitalized for AHF presenting with clinical evidence of fluid overload. The study will evaluate natriuresis at 24 and 48 hours following intravenous acetazolamide administration in patients with persistent congestion despite treatment with intravenous furosemide and an SGLT2i. Upon admission, all patients will receive intravenous loop diuretics according to current European guideline recommendations. For those not previously treated with an SGLT2i, therapy will be initiated within the first 24 hours. Congestion will be reassessed 24 hours after combined loop diuretic and SGLT2i therapy. In line with the ADVOR trial, patients with persistent congestion (ADVOR score > 1) will receive intravenous acetazolamide (500 mg once daily) for up to two consecutive days.

During hospitalization and follow-up, participants will be encouraged to limit their daily dietary sodium and fluid intake to 3 g and 1500 ml, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted for acute heart failure and ≥ 1 clinical sign of volume overload (edema, ascites, or pleural effusion).
* NTproBNP levels >1000 pg/mL or BNP >250 ng/mL on admission.
* Under treatment with furosemide and iSGLT2 according to European guidelines and indication of association of another diuretic due to residual congestion data defined by ADVOR SCORE>1.

Exclusion Criteria:

* Systolic blood pressure <90 mmHg or mean arterial pressure < 65 mmHg.
* Maintenance treatment with acetazolamide/ Treatment with acetazolamide in the month prior to inclusion in the study.
* Anticipated need for intravenous inotropes, vasopressors or nitroprusside during the study.
* Contraindication to ISGLT2.
* Type 1 diabetes mellitus
* GFR < 20 ml/min/m2 or renal replacement therapy/ultrafiltration at any time prior to the study.
* Anticipated exposure to nephrotoxic agents, such as iodinated contrast during admission.
* Concurrent diagnosis of acute coronary syndrome.
* History of congenital heart disease requiring surgical correction.
* History of cardiac transplantation and/or ventricular assist device.
* Pregnant or breastfeeding patients.
* Inability to adequately collect diuresis.
* Serum potassium less than 3.5 mEq/L.
* Venous pH <7.30
* Severe aortic stenosis or obstructive hypertrophic cardiomyopathy.
* Sulfonamide allergy, liver cirrhosis, renal lithiasis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted for heart failure with persistent findings of residual congestion who meet the inclusion criteria and none of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in natriuresis 24 hours after acetazolamide | 24 hours
  Change in natriuresis (mmol) 24 hours after acetazolamide association to medical treatment recommended by the guidelines (furosemide and ISGLT2).

SECONDARY OUTCOMES:
Increase in diuresis 24 hours after acetazolamide administration | 24 hours
  Increase in diuresis 24 hours after acetazolamide administration (liters)
Weight difference 24 hours after acetazolamide administration | 24 hours
  Weight difference 24 hours after acetazolamide administration (Kg)
Difference in congestion score 24 hours after acetazolamide administration. | 24 hours
  Difference in congestion score 24 hours after acetazolamide administration using ADVOR congestion score. It is a 0-10 scale used in the ADVOR trial to objectively quantify volume overload in acute heart failure, based on three components: peripheral edema scored from 0 to 4 points, pleural effusion from 0 to 3 points, and ascites from 0 to 3 points. A total score of 0 represents the absence of measurable congestion, while the maximum of 10 indicates severe, multisite fluid accumulation. Higher ADVOR scores reflect more severe congestion.
Difference in ultrasound measurement of Inferior Vena Cava 24 hours after acetazolamide administration. | 24 hours
  Difference in inferior vena cava size (mm) assessed by ultrasound, he IVC is visualized in the subcostal long-axis view, and its diameter is measured about 1-2 cm from its junction with the right atrium, 24 hours after acetazolamide administration
Change in natriuresis 48 hours after acetazolamide administration | 48 hours
  Change in natriuresis 48 hours after acetazolamide administration
Change in diuresis 48 hours after acetazolamide administration | 48 hours
  Change in diuresis 48 hours after acetazolamide administration
Weight difference 48 hours after acetazolamide administration | 48 hours
  Weight difference 48 hours after acetazolamide administration
Difference in congestion score 48 hours after acetazolamide administration. | 48 hours
  Difference in congestion score 48 hours after acetazolamide administration using ADVOR congestion score. It is a 0-10 scale used in the ADVOR trial to objectively quantify volume overload in acute heart failure, based on three components: peripheral edema scored from 0 to 4 points, pleural effusion from 0 to 3 points, and ascites from 0 to 3 points. A total score of 0 represents the absence of measurable congestion, while the maximum of 10 indicates severe, multisite fluid accumulation. Higher ADVOR scores reflect more severe congestion.
Difference in ultrasound measurement of Inferior Vena Cava 48 hours after acetazolamide administration. | 48 hours
  Difference in inferior vena cava size (mm) assessed by ultrasound. The IVC is visualized in the subcostal long-axis view, and its diameter is measured about 1-2 cm from its junction with the right atrium, 48 hours after acetazolamide administration
Change in Vexus score 24 hours after acetazolamide administration. | 24 h post acetazolamide administration
  Vexus score: The VExUS score (Venous Excess Ultrasound Score) is an ultrasound-based grading system used to assess systemic venous congestion by integrating measurements of the inferior vena cava (IVC) and Doppler patterns of key abdominal veins: the hepatic vein, portal vein, and intrarenal vein. A dilated IVC combined with progressively abnormal venous Doppler waveforms indicates increasing venous congestion. VExUS is typically graded from 0 to 3, where Grade 0 represents no significant congestion and Grade 3 indicates severe venous congestion with markedly abnormal waveforms across multiple veins. Higher VExUS correlates with worse outcomes.

OTHER OUTCOMES:
Changes in renal function 24 hours after acetazolamide administration. | 24 hours
  Changes in renal function assessed by differences in serum creatinine (mg/dL)24 hours after acetazolamide administration.
Ionic (potassium (mmol/L) changes | 24 hours
  Ionic (potassium (mmol/L) changes 24 hours after acetazolamide
chloride (mmol/L) changes 24 hours after acetazolamide administration | 24 hours
  chloride (mmol/L) changes 24 hours after acetazolamide
bicarbonate (mmol/L) changes 24 hours after acetazolamide administration | 24 hours
  bicarbonate (mmol/L) changes 24 hours after acetazolamide administration
Changes in systolic blood pressure 24 hours after administration of acetazolamide | 24 hours
  Changes in systolic blood pressure 24 hours after administration of acetazolamide (mmHg)
Changes in renal function 48 hours after acetazolamide administration | 48 hours
  Changes in renal function assessed by differences in serum creatinine (mg/dL) 48 hours after acetazolamide administration.
Ionic (potassium (mmol/L) changes 48 hours after acetazolamide administration | 48 hours
  Ionic (potassium (mmol/L) changes 48 hours after acetazolamide
Chloride (mmol/L) changes 48 hours after acetazolamide administration | 48 hours
  Chloride (mmol/L) changes 48 hours after acetazolamide
Bicarbonate (mmol/L) changes 48 hours after acetazolamide administration | 48 hours
  Bicarbonate (mmol/L) changes 48 hours after acetazolamide administration
Changes in systolic blood pressure 48 hours after administration of acetazolamide | 48 hours
  Changes in systolic syblood pressure 48 hours after administration of acetazolamide (mmHg)
Change in Vexus score 48 hours after acetazolamide administration. | 48 hours post acetazolamide administration
  Vexus score: The VExUS score (Venous Excess Ultrasound Score) is an ultrasound-based grading system used to assess systemic venous congestion by integrating measurements of the inferior vena cava (IVC) and Doppler patterns of key abdominal veins: the hepatic vein, portal vein, and intrarenal vein. A dilated IVC combined with progressively abnormal venous Doppler waveforms indicates increasing venous congestion. VExUS is typically graded from 0 to 3, where Grade 0 represents no significant congestion and Grade 3 indicates severe venous congestion with markedly abnormal waveforms across multiple veins. Higher VExUS correlates with worse outcomes.
Change in lung B-lines 24 hours after acetazolamide administration | 24 hours
  Change in the number of lung zones with B-lines assessed by lung ultrasound 24 hours after acetazolamide administration. The 8-zone lung ultrasound method evaluates pulmonary congestion by scanning four zones on each hemithorax (anterior and lateral, each divided into upper and lower fields). In each zone, the operator assesses the pleural line and counts B-lines. A zone is considered positive if it contains more than three B-lines
Change in lung B-lines 48 hours after acetazolamide administration | 48 hours
  Change in the number of lung zones with B-lines assessed by lung ultrasound 48 hours after acetazolamide administration. The 8-zone lung ultrasound method evaluates pulmonary congestion by scanning four zones on each hemithorax (anterior and lateral, each divided into upper and lower fields). In each zone, the operator assesses the pleural line and counts B-lines. A zone is considered positive if it contains more than three B-lines

CONTACTS AND LOCATIONS:
Locations (1):
- Julia González González, Madrid, Spain